CLINICAL TRIAL: NCT00004008
Title: A Phase II Trial of Bryostatin 1 in Ovarian Cancer Administered by Weekly 24 Hour Intravenous Infusion
Brief Title: Bryostatin 1 in Treating Patients With Ovarian Epithelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Glasgow (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CRC-PHASE-II-PH2/039; CDR0000067219 (Registry Identifier: PDQ (Physician Data Query)); NCI-T99-0027
Record Dates: First submitted 1999-11-01; First posted 2003-05-08 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 1999-11

CONDITIONS: Ovarian Cancer
Keywords: stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — bryostatin 1

INTERVENTIONS:
Drug: bryostatin 1

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of bryostatin 1 in treating patients who have ovarian epithelial cancer that has not responded to previous chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the antitumor activity and toxicity of bryostatin 1 in patients with platinum resistant ovarian epithelial cancer.
* Determine the response rate in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive bryostatin 1 IV over 24 hours. Treatment repeats weekly for 8 courses in the absence of disease progression or unacceptable toxicity. Patients achieving stable or regressive disease may receive additional treatment.

Patients are followed for at least 4 weeks after treatment, then every 3 months.

PROJECTED ACCRUAL: A total of 14-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven ovarian epithelial cancer

  * Progressive disease during or after completion of at least one platinum based chemotherapy regimen
* Bidimensionally measurable disease

  * At least 2 cm by x-ray, CT scan, or ultrasound
* No active, symptomatic brain metastases (e.g., cerebral edema and/or progressive tumor growth)

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* WHO 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Hemoglobin at least 10 g/dL
* WBC at least 4,000/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin no greater than 1.7 mg/dL
* AST/ALT no greater than 2.5 times upper limit of normal (ULN) (no greater than 5 times ULN if liver metastases present)

Renal:

* Creatinine no greater than 1.4 mg/dL

Other:

* No active, uncontrolled infection
* No nonmalignant systemic disease which would increase risk to patient
* No other malignancies within the past 5 years except curatively treated basal or squamous cell skin cancer or carcinoma in situ of the cervix
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks since nitrosoureas or mitomycin) and recovered
* No more than 2 prior multidrug chemotherapy regimens
* No more than 1 prior single agent chemotherapy regimen

Endocrine therapy:

* At least 4 weeks since prior endocrine therapy and recovered
* No concurrent steroids
* Concurrent hormone replacement therapy allowed

Radiotherapy:

* At least 4 weeks since prior radiotherapy (excluding palliative therapy) and recovered
* No concurrent radiotherapy

Surgery:

* At least 4 weeks since prior major thoracic or abdominal surgery

Other:

* No other concurrent anticancer therapy or investigational drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-07; Study Completion 2003-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Jayson, MD, Study Chair — The Christie NHS Foundation Trust
Locations (4):
- United Kingdom (4):
  - Christie Hospital N.H.S. Trust, Manchester, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Weston Park Hospital, Sheffield, England
  - Royal Infirmary, Glasgow, Scotland